CLINICAL TRIAL: NCT01914341
Title: Short-term Effects of Live Pentatonic Music on Physiological Parameters in Newborns Infants
Brief Title: Short Term Effects of Live Music in Newborn Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ARCIM_MTN04
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Newborn Infant
Keywords: Infant; Newborn; Music
MeSH Terms: interventions — Music Therapy

ARMS (2):
- Music (Experimental): pentatonic live music
  Interventions: Other: Music
- control (No Intervention): no intervention

INTERVENTIONS:
Other: Music — Live music played on the pentatonically tuned children's harp
  Arms: Music

SUMMARY:
The purpose of this study is to determine the effects of live music on physiological parameters in newborn infants. The mother is asked about the effects of music on her own and the child's wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 35 weeks
* signed informed consent of the parents
* positive proof of hearing ability (TEOAE, transitory evoked otoacoustic emission)
* positive 10-minute Apgar-Score > 7

Exclusion Criteria:

* Heart defect or known cardiac arrhythmia
* other diseases of the preterm and newborn period (including infections and chromosomal aberrations)
* participation in other studies

Min Age: 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
heartrate | physiological parameters are measured twice over a period of 45 minutes

SECONDARY OUTCOMES:
Oxygen saturation | physiological parameters are measured twice over a period of 45 minutes.
Breathing rate | physiological parameters are measured twice over a period of 45 minutes
Apnoea > 4 sec per hour | physiological parameters are measured twice over a period of 45 minutes
Bradycardia < 80 bpm/h | physiological parameters are measured twice over a period of 45 minutes
Tachycardia > 200 bmp/h | physiological parameters are measured twice over a period of 45 minutes
heart rate variability-parameters (HRV) | physiological parameters are measured twice over a period of 45 minutes
  RMSS (root mean square of successive differences) SDNN (standard deviation of normal to normal intervals) pNN50 (the proportion of NN50 (the number of pairs of successive NNs that differ by more than 50 ms) divided by total number of NNs) LF/HF (low frequency/high frequency)
Perfusion Index (PI) | physiological parameters are measured twice over a period of 45 minutes
Pulse-Transit-Time (PTT) | physiological parameters are measured twice over a period of 45 minutes
State Trait Anxiety Inventory | Questionnaires are filled in by the child's mother before and after the music intervention respectively no intervention (during the first and during the last 15 minutes of the physiological measurement).
State of the child | Questionnaires are filled in by the child's mother before and after the music intervention respectively no intervention (during the first and during the last 15 minutes of the physiological measurement).
Additional music questions | The additional music questions are filled in by the child's mother after the music intervention (during the15 minutes directly after the music intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Principal Investigator — ARCIM-Institute; University Hospital Tuebingen
Locations (1):
- Filderklinik, Filderstadt, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Arnon S, Shapsa A, Forman L, Regev R, Bauer S, Litmanovitz I, Dolfin T. Live music is beneficial to preterm infants in the neonatal intensive care unit environment. Birth. 2006 Jun;33(2):131-6. doi: 10.1111/j.0730-7659.2006.00090.x. PMID 16732778
- [Background] Bo LK, Callaghan P. Soothing pain-elicited distress in Chinese neonates. Pediatrics. 2000 Apr;105(4):E49. doi: 10.1542/peds.105.4.e49. PMID 10742370
- [Background] Standley JM. A meta-analysis of the efficacy of music therapy for premature infants. J Pediatr Nurs. 2002 Apr;17(2):107-13. doi: 10.1053/jpdn.2002.124128. PMID 12029604